CLINICAL TRIAL: NCT03656445
Title: Multiple Intravenous Tranexamic Acid Doses Can Reduce Postoperative Blood Loss and Improve the Functional Outcome in Total Knee Arthroplasty Without Tourniquet: a Randomized Controlled Study
Brief Title: Tranexamic Acid in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Tzatzairis Themistoklis, Principal investigator Dr. Tzatzairis Themistoklis, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 546a - 26/10/2015
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Osteo Arthritis Knee
Keywords: total knee arthroplasty; tranexamic acid; without tourniquet; blood loss; function; multiple doses
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - Tranexamic Acid (Active Comparator): 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, 10 minutes before incision, administered during the induction of the anesthesia
  Interventions: Drug: Tranexamic Acid
- Group B - Tranexamic Acid (Active Comparator): 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, 10 minutes before incision and an additional dose of IV TXA (15mg/kg) in 100-ml normal saline 3 hours after skin incision
  Interventions: Drug: Tranexamic Acid
- Group C - Tranexamic Acid (Active Comparator): 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, before incision and two additional doses of IV TXA (15mg/kg) in 100-ml normal saline 3 and 6 hours after skin incision respectively
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, 10 minutes before incision, administered during the induction of the anesthesia
  Other Names: Transamin; Cyklokapron
  Arms: Group A - Tranexamic Acid
Drug: Tranexamic Acid — 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, 10 minutes before incision and an additional dose of IV TXA (15mg/kg) in 100-ml normal saline 3 hours after skin incision
  Other Names: Transamin; Cyklokapron
  Arms: Group B - Tranexamic Acid
Drug: Tranexamic Acid — 1 dose of IV TXA (15mg/kg) in 100-ml normal saline, before incision and two additional doses of IV TXA (15mg/kg) in 100-ml normal saline 3 and 6 hours after skin incision respectivel
  Other Names: Transamin; Cyklokapron
  Arms: Group C - Tranexamic Acid

SUMMARY:
Multiple intravenous Tranexamic Acid doses can reduce postoperative blood loss and improve the functional outcome in total knee arthroplasty without tourniquet: a randomized controlled study.

DETAILED DESCRIPTION:
A total of 180 patients undergoing TKA for knee osteoarthritis were stratified in three equal groups. All surgeries were performed under spinal anesthesia, without tourniquet and patients should be in agreement with the established inclusion/exclusion criteria. Group A (60 patients) received 1g of IV TXA, Group B (60 patients) received an additional dose of IV TXA and Group C (60 patients) received three doses of IV TXA. The measured outcomes were the Hemoglobin (Hb) decrease, the transfusion rate, the functional, quality of life (QoL) and pain assessment based on their corresponding scoring system.

ELIGIBILITY:
Inclusion Criteria:

1. varus deformity less than 10o
2. lack of extension not more than 10o
3. flexion of at least 90o.

Exclusion Criteria:

1. uncontrolled medical diseases/comorbidities
2. allergy and/or hypersensitivity to TXA
3. a known history of thromboembolic disease, cardiovascular disease
4. coronary or vascular stent placed within the past 12 months
5. cerebral vascular disease (a history of stroke)
6. subarachnoid hemorrhage
7. preoperative coagulopathy (a platelet [PLT] count <150,000/mm3 or an international normalized ratio greater than 1.5
8. preoperative renal or hepatic dysfunction
9. retinal vein or artery occlusion
10. patients with anemia (<12 g/dL for female, <13 g/dL for male)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
hemoglobin change | 1st,2nd and 4th post-operative day
  Hemoglobin decrease/change during the four post-operative days
Blood loss | 24 hours
  calculated total blood loss (TBL) the 1st post-op day
Blood loss | 48 hours
  calculated total blood loss (TBL) the 2nd post-op day
Blood loss | 96 hours
  calculated total blood loss (TBL) the 4th post-op day
Platelet count change | 24 hours, 48 hours, 96 hours
  Platelet count increase/decrease/change during the 1st,2nd and 4th day
Need for trasfussion | 24 hours
  Transfussion rate/quantity in 1st post-op day
Need for trasfussion | 48 hours
  Transfussion rate/quantity in 2nd post-op day
Need for trasfussion | 96 hours
  Transfussion rate/quantity in 3rd post-op day

SECONDARY OUTCOMES:
Knee Society Score (KSS) KSS | 2nd and 4th post op days + 6th week and 12th week
  Change in this Score which is an objective scoring system to rate the knee and patient's functional abilities such as walking and stair climbing before and after TKA. Maximum score is 100 (best functionality) and lowest score is 0 (worst functionality)
Function Knee Society Score | 2nd and 4th post op days + 6th week and 12th week
  Change in this score which utilizes walking distance and stair climbing as the main parameters, with deduction for the use of a walking aid. Maximum score is 100 (best functionality) and lowest score is 0 (worst functionality)
EuroQol | 2nd and 4th post op days + 6th week and 12th week
  Changes in this score which is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. Crosswalk value sets for the EQ-5D-5L has been used to asses the results into numbers. Maximum score is 1 (which means best quality of life) and the lowest is -0.594(which means the worst quality of life)
VAS pain (analogue pain scale) | 2nd and 4th post op days + 6th week and 12th week
  The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10 [100-mm scale])

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clinics in geriatric medicine. Aug 2010;26(3):355-369. 2. Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. British medical bulletin. 2013;105:185-199. 3. Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. The Journal of bone and joint surgery. American volume. Apr 2007;89(4):780-785. 4. Bourne RB, McCalden RW, MacDonald SJ, Mokete L, Guerin J. Influence of patient factors on TKA outcomes at 5 to 11 years followup. Clinical orthopaedics and related research. Nov 2007;464:27-31. 5. Anderson JG, Wixson RL, Tsai D, Stulberg SD, Chang RW. Functional outcome and patient satisfaction in total knee patients over the age of 75. The Journal of arthroplasty. Oct 1996;11(7):831-840. 6. Mulhall KJ, Ghomrawi HM, Bershadsky B, Saleh KJ. Functional improvement after total knee arthroplasty revision: new observations on the dimensional nature of outcome. Journal of orthopaedic surgery and research. Dec 07 2007;2:25. 7. Saleh KJ, Dykes DC, Tweedie RL, et al. Functional outcome after total knee arthroplasty revision: a meta-analysis. The Journal of arthroplasty. Dec 2002;17(8):967-977. 8. Sikorski JM. Alignment in total knee replacement. The Journal of bone and joint surgery. British volume. Sep 2008;90(9):1121-1127. 9. Blumberg N. Allogeneic transfusion and infection: economic and clinical implications. Semin Hematol. 1997/07// 1997;34(3 Suppl 2):34-40. 10. Vamvakas EC, Blajchman MA. Transfusion-related mortality: the ongoing risks of allogeneic blood transfusion and the available strategies for their prevention. Blood. Apr 09 2009;113(15):3406-3417. 11. Berry DJ, Bozic KJ. Current practice patterns in primary hip and knee arthroplasty among members of the American Association of Hip and Knee Surgeons. The Journal of arthroplasty. Sep 2010;25(6 Suppl):2-4. 12. Themistoklis T, Theodosia V, Konstantinos K, Georgios DI. Perioperative blood management strategies for patients undergoing total knee replacement: Where do we stand now? World journal of orthopedics. Jun 18 2017;8(6):441-454. 13. Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. Journal of orthopaedic surgery and research. 2014;9:13-13. 14. Zhang Q, Dong J, Gong K, Li X, Zheng S, Wen T. [Effects of Tourniquet Use on Perioperative Outcome in Total Knee Arthroplasty]. Zhongguo xiu fu chong jian wai ke za zhi = Zhongguo xiufu chongjian waike zazhi = Chinese journal of reparative and reconstructive surgery. Apr 2016;30(4):421-425. 15. Du Z, Liu P, Zhang Y, Li D, Li M. [Effect of tourniquet on perioperative blood loss and short-term effectiveness in total knee arthroplasty]. Zhongguo xiu fu chong jian wai ke za zhi = Zhongguo xiufu chongjian waike zazhi = Chinese journal of reparative and reconstructive surgery. Nov 2013;27(11):1318-1323. 16. Li X, Yin L, Chen ZY, et al. The effect of tourniquet use in total knee arthroplasty: grading the evidence through an updated meta-analysis of randomized, controlled trials. European journal of orthopaedic surgery & traumatology : orthopedie traumatologie. Aug 2014;24(6):973-986. 17. Tetro AM, Rudan JF. The effects of a pneumatic tourniquet on blood loss in total knee arthroplasty. Canadian journal of surgery. Journal canadien de chirurgie. Feb 2001;44(1):33-38.